CLINICAL TRIAL: NCT05323344
Title: Metacognitive Therapy and Neuro-physiotherapy as a Treatment for Functional Movement Disorders - a Randomized, Observer-blinded Feasibility Trial
Brief Title: Metacognitive Therapy and Neuro-physiotherapy as a Treatment for Functional Movement Disorders
Acronym: ReMAP-FMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Anne Weißbach, Principle Investigator, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WE5919/4-1
Record Dates: First submitted 2022-03-21; First posted 2022-04-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Conversion Disorder
Keywords: functional movement disorders; feasibility study; Physiotherapy; Metacognitive behavioral therapy
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: Feasibility study
Who Masked: Outcomes Assessor
Masking Description: Blinded video rating for primary endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-physiotherapy (Active Comparator): In intervention group I, patients will receive a one hour session of special Neuro-physiotherapy (NPT) twice per week with a total of 20 sessions over 10 weeks. In addition, patients will be instructed to a home-based training, so that they continue their training in between sessions and after completion of the 10 weeks intervention. NPT is designed to target the abnormal movements. It is based on previously established consensus recommendations and feasibility for a short (5 days) intervention was already tested. Adapted from Nielsen et al., each of our NPT sessions will include patient education, movement retraining and development of a self-management plan.
  Interventions: Other: Neuro-physiotherapy
- Combination of metacognitive therapy and Neuro-physiotherapy (Active Comparator): In intervention group II, patients will be treated for 10 weeks by a combination of Metacognitive behavioral therapy (MCT) and Neuro-physiotherapy (NPT) (1 hour MCT and 1 hour NPT per week with a total of 20 treatment sessions over 10 weeks). The key feature during MCT sessions will be based on an attention training technique (ATT), which prevents or interrupts self-focused attention and reduces the overall level of preoccupation with the FMD. Patients will receive at least three competing sounds. Patients will be asked to practice the training with their eyes open and focused on a visual fixation point. Patients' self-reliance will be strengthened by an individualized cognitive self-training explained and practiced with the MCT therapist including an audio tape of the ATT training. This should be continued daily at home in between sessions and after completion of the 10 weeks intervention. Self-training will be documented in a daily training diary.
  Interventions: Other: Combination of metacognitive behavioral therapy and Neuro-physiotherapy

INTERVENTIONS:
Other: Neuro-physiotherapy — Neuro-Physiotherapy will be done in Intervention group I
  Arms: Neuro-physiotherapy
Other: Combination of metacognitive behavioral therapy and Neuro-physiotherapy — Combination of metacognitive behavioral therapy and Neuro-physiotherapy will be done in intervention group II
  Arms: Combination of metacognitive therapy and Neuro-physiotherapy

SUMMARY:
Patients with functional movement disorders (FMD) present with abnormal movements incompatible with symptoms of well-defined neurological disorders and are not associated with structural abnormality of the nervous system. FMD are very common. However, the pattern of care of these patients is highly inconsistent and most patients feel dissatisfied with the treatment they receive. One reason for this unsatisfactory scenario is that there are no generally accepted therapeutic guidelines for FMD.

Therefore, treatment strategies are urgently needed. Recent neurophysiological studies suggest common underlying disease mechanism across FMD patients, particularly abnormal allocation of attentional resources. Conceptually, this calls for therapeutic approaches, in which attention re-focusing is trained. In this respect, neuro-physiotherapy (NPT) is based on the physical movement retraining by demonstrating that normal movement is possible, to facilitate patients' confidence into the own movement capacity. Based on the current literature, the investigators suggest that NPT is a feasible and effective treatment options in FMD population. However, the proportion of patients fully accepting and improving from NPT was limited. FMD patients might be more receptive to NPT if additional specialized psychotherapy approaches, e.g., metacognitive therapy (MCT) is offered. MCT focusses on patients believes about their own mind and cognition (metacognition). It explains how dysfunctional patterns of thinking and self-awareness can lead to and maintain FMD and in particular trains patients to consciously (re-)focus their attention away from unpleasant or disturbing mental processes. Thus, the investigators aim to analyze, in addition to NPT only, the feasibility and treatment efficacy of a combination of NPT and MCT.

The investigators will apply therapy frequently (2 times 1 hour sessions per week over 10 weeks) and patients will be instructed for an additional home-based training. Effectiveness will be analyzed up to 12 month after the intervention by validated, FMD-specific, blinded video ratings.

Importantly, FMD patients have been shown to have the potential for a full recovery if sufficient treatment is applied. Therefore, the therapeutic approaches of the clinical feasibility trial, if successful, are expected to have immediate and strong impact on the care of FMD patients including an improvement in quality of life, and to reduce health care system burdens.

DETAILED DESCRIPTION:
Trial Design The proposed clinical feasibility pilot study contains two intervention groups. Patients with functional movement disorders (FMD) will be randomized into the two groups. Patients of the intervention group I will receive 10 weeks neuro-physiotherapy (NPT) and patients of the intervention group II a combination of NPT and metacognitive therapy (MCT).

Frequency and Scope of Trial Visits At a screening visit before participation in the clinical trial all patients will be assessed for eligibility by applying the inclusion and exclusion criteria and will be provided with information to obtain informed consent. If eligible, patients are randomized to the two different groups. At baseline examination, social demographic information (age, gender, education, family status etc.) and medical history (age at onset, disease duration, potential triggers, comorbidities, previous therapies etc.) are obtained. At baseline, immediately after completion of the intervention and at three, six and 12 months follow-up visits the investigators will use a standardized video protocol that ensures consistent examination of the movement disorder according to a standardized video-guided instruction protocol. It allows a blinded, objective video rating of patients' symptoms at all five study visits by the investigators that will stay blinded to the treatment status of the patient. Both have extensive experience in design, conduction and analysis of movement disorders video ratings. They will rate the severity of symptoms by applying clinical rating scales and questionnaires for patients with functional movement disorders. The baseline visit will take two hours and the post-interventional as well as follow-up visits will each last one hour.

Medical Problem and Relevance Patients with FMD present with different abnormal movements such as functional tremor, dystonia, myoclonus, or gait disorders and often also other symptoms and signs suggesting the involvement of the nervous system. FMD are incompatible with symptoms and signs of well-defined neurological disorders and are not associated with structural abnormality of the nervous system. Importantly, FMD disorders can reliably be diagnosed clinically on the basis of characteristic signs including incongruency of symptoms regarding anatomy and physiology, variable phenomenology, attention dependency, i.e. increased distractibility, entrainment and other specific signs, for instance, Hoover's sign. Thus, FMD is not a diagnosis of exclusion. Although FMD were referred to as "psychogenic" or "conversion movement disorder" suggesting psychopathology as a pre-requisite, a high percentage of patients in fact do not have psychiatric comorbidities.

The level of distress, disability and chronification of symptoms in patients with FMD is comparable to or even higher than that in patients with defined neurological disorders. FMDs are very common and along with other disorders in the spectrum of functional neurological disorders (FND), account for up to one-third of new referrals seen in neurology clinics. Their prevalence in private neurological practices is about 16% and almost as high as patients with headaches (19%) or epilepsy (14%). FMDs account for up to 20% of patients seen in movement disorders clinics. However, the pattern of care of these patients is highly inconsistent and most patients feel dissatisfied with the treatment they receive.

One reason for this unsatisfactory scenario that is also severely affecting the German healthcare system, is that there are no generally accepted therapeutic guidelines for FND patients. Often, patients are referred from one specialist to the other with neither neurologist nor psychiatrist taking on the long-term care for these patients due to a lack of validated treatment strategies. Patients typically seek advice from different specialists and often receive unnecessary, cost intensive diagnostic procedures that might be associated with complications. This leads to further referrals, unnecessary use of valuable health care system resources and secondary iatrogenic morbidity. The Scottish Neurological Symptom Study showed that patients suffering from FND create direct health care cost of about £11.3 million per year in Scotland. A study from the USA estimated the direct healthcare cost of FND patients in the USA of about $256 billion. In comparison to other neurological disorders, FND patients demand not only significantly more primary, specialty and emergency care visits, but also in- and outpatient clinic administrations.

Therefore, treatment strategies meeting FMD patients' needs are urgently needed. However, finding effective treatment is complicated by the fact that clinical symptoms of FMD are highly heterogeneous. Interestingly, recent neurophysiological studies suggest common underlying disease mechanism across FMD patients. For instance, in a temporal discrimination paradigm, FMD patients had reduced drift rates pointing towards a generalized deficit in information processing. In addition, FMD patients showed a significant reduction of physiological attenuation of self-generated perceptual stimuli reflecting an altered sense of agency, probably as a consequence of aberrant allocation of attentional recourses, which may also explain why voluntary movements are not experienced as such. Conceptually, this calls for therapeutic approaches, in which attention re-focusing is trained. In this respect, MCT and NPT are promising treatment options. MCT, as a form of cognitive behavioral therapy, focusses on patients believes about their own mind and cognition (metacognition). It explains how dysfunctional patterns of thinking and self-awareness can lead to and maintain FMDs and trains patients to consciously (re)-focus their attention away from unpleasant or disturbing mental processes. It has been successfully established in a pilot study conducted at the investigators' study site (University Clinic Schleswig-Holstein = UKSH) for the treatment of patients with Gilles de la Tourette syndrome. NPT is based on physical movement retraining by demonstrating that normal movement is (at least in parts) possible, to facilitate patients' confidence into their own movement capacity.

Importantly, FMD patients have the potential for a full recovery if sufficient treatment is applied. Therefore, the therapeutic approaches of the clinical trial, if successful, are expected to have immediate and strong impact on the care of FMD patients including an improvement in quality of life and to reduce health care system burdens. The latter is particularly relevant in the current coronavirus disease 19 (COVID-19) pandemic given that the incidence of FMD is known to rise with social crises. This is, at least partly, explained by the fact that fear and uncertainty are known to increase the incidence of neuropsychiatric disorders including FMDs.

Justification of Design Aspects Results of the proposed feasibility pilot study will provide important information on NPT and combined NPT/MCT effect size for the power and sample size calculations of a subsequently planned multicenter confirmatory trial. Moreover, patients' acceptance of interventions will be investigated in the proposed feasibility study. According to patients' feedback, adaptation of the interventions for a subsequent confirmatory trial will be possible.

Proposed Sample Size / Power Calculations Sample size was calculated with the aim to ensure that the effect of the interventions can be estimated with sufficient precision. For this purpose, the effect is based on the individual change in motor scores between baseline and after twelve months. Based on data from the only study with published individual patient scores (PMDRS) before and after cognitive behavioral therapy, a decrease of scores after the intervention can be expected with a mean(delta) of -26.87 and SD(delta) of 18.58. From this, it can be estimated that a sample size of 19 patients is sufficient to ensure that the 95% confidence interval of this mean delta is not wider than +/- 50% of the SD of the baseline scores, meaning that a change in pre- to post-interventional scores can be estimated with +/- 0.5 SD accuracy with a probability of 95%. Given that effects are to be estimated in both treatment groups and compared with each other, 19 patients need to be available for analysis in every group. Sample size calculation was performed using nQuery.

Compliance / Rate of Loss to Follow-Up The investigators identified six studies using physiotherapy and seven studies applying psychotherapy that reported exclusion rates during assessment for eligibility and drop-out rates from follow-up visits. Due to this information, the investigators calculated a mean rate of loss to follow-up of about 19% and exclusion rates during assessment for eligibility of 33%. Therefore, the investigators plan to enroll 61 patients and randomize 46 patients over the two groups. According to the drop-out rates, this will leave us with 19 patients per group to be analyzed

Statistical Analysis All analyzes will be performed for descriptive purposes. For primary and secondary endpoints, differences between intervention groups will be estimated with accompanying confidence intervals for every follow-up time. For all remaining variables, location and variation parameters will be estimated depending on their measurement scale. Analyzes of primary and secondary endpoints will be performed both in intention-to-treat as well as per-protocol populations.

In this feasibility study, no missing values will be imputed, and no interim analyzes are planned.

The results of this feasibility study will be used for effect size calculations for a subsequent multicenter confirmatory trial. All statistical analyzes were and will be done at the Institute of Medical Biometry and Statistics, University of Lübeck.

Quality Assurance, Safety, Monitoring and Data Reviewing Measures of quality assurance and safety will be done by a highly qualified clinical research associate at the Center for Clinical Trials Lübeck (ZKS). They will include clinical onsite risk-based monitoring according to ICH-GCP guideline (E6) and written standard operating procedures (SOPs) of the ZKS network to ensure patients' rights, patients' security and reliability of trial results. According to those SOPs, monitoring activities will be defined in a monitoring manual before starting the trial.

To initiate the study, the two trial sites will be visited by a clinical research associate of the ZKS Lübeck. During the ongoing trial, sites will be visited again at least two times to check informed consents and defined key data of all patients. Due to the low risk of the two interventions patient files will be randomly screened for adverse and serious adverse events. Within the frame of source data verification (SVD) during the trial, case report forms, patients' self-questionnaires and clinical ratings will be checked within a defined number of patients during the two onsite visits. At the end of the clinical trial, the two sites will be closed by a close-out visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinically established diagnosis of functional movement disorders (FMD) according to the revised Fahn-Williams criteria. Patients with FMD with different phenomenology, i.e. patients with functional myoclonus, dystonia, tremor and functional gait disorders will be included to guarantee generalizability and representativeness of this heterogeneous disorder.

Exclusion Criteria:

* Significant major neuropsychiatric/neurological disorder
* medical illness with known central nervous system consequences,
* acute unstable psychiatric diseases,
* pain disorders,
* paroxysmal FMD,
* isolated functional paresis,
* inability to read and speak German,
* age < 18 years. Children with FMD are excluded because they would require age-adjusted assessment and tailored treatment in a specialized neuropediatric unit.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Score on the Simplified Functional Movement Disorders Rating Scale (S-FMDRS) between baseline and up to one week after intervention | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician-rated, rating scale for functional motor symptoms; used for blinded video rating

SECONDARY OUTCOMES:
Changes in Score on the Psychogenic movement disorders rating scale (PMDRS) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician-rated, rating scale for functional motor symptoms; used for blinded video rating
Changes in Score on the Clinical Global Impression-Severity and Improvement (CGI-S and CGI-I) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician- and patient-rated, general symptom severity and improvement
Changes in Score on the Clinical Global Impression (CGI) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician- and patient-rated, general symptom severity and improvement
Changes in Score on the Short Form Health Survey-36 (SF-36) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire
Changes in Score on the Fatigue Assessment Scale | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire
Changes in Score on the Beck Depression Inventory-II (BDI-II) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire on depression severity
Changes in Score on the Hospital Anxiety and Depression Scale (HADS) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire; anxiety and depression severity
Changes in Score on the The Meta-cognition questionnaire | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire on thinking about patients own cognition
Changes in Score on the Positive and Negative Effects of Psychotherapy Scale (PANEPS) | up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire on treatment acceptance
Changes in Score on the World Health Quality of Life assessment (WHOQOL) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire; global quality of life
Changes in Score on the Client Sociodemographic and Service Receipt Inventory (CSSRI) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire
Changes in Score on the Clinical rating scale for tremor | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician-rated, tremor severity, rated by blinded video rating
Changes in Score on the Timed up and go test | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician-rated, mobility and balance, rated by blinded video rating
Changes in Score on the "Tinetti test" | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician-rated, risk of falling, rated by blinded video rating
Changes in Score on the Berg balance test | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician-rated, balance, rated by blinded video rating
Changes in Score on the Questionnaire for functional movement disorders | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Clinician and self-rated patients questionnaire, subjective complaints and impacts of functional movement disorders
Changes in Score on the Bochum Change Questionnaire 2000 | up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire; direct measurement of change in psychotherapy
Changes in Score on the Work and Social Adjustment Scale (WSAS) | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Self-rated patients questionnaire

OTHER OUTCOMES:
Transcranial magnetic stimulation | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  Dual-pulse paradigm investigating connectivity between the primary motor cortex and the temporal-parietal junction
Magnetic resonance imaging (DTI) | baseline, 3, 12 month follow-up
  Diffusion Tensor Imaging sequence of the entire brain
Magnetic resonance imaging (Resting State) | baseline, 3, 12 month follow-up
  Magnetic resonance imaging of the entire brain while the patient is at rest
Magnetic resonance imaging (T1) | baseline, 3, 12 month follow-up
  high-resolution T1-weighted sequence of the entire brain
Motor metacognition task | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  The metacognition motor task will be done on an electronic writing pad. The patients are instructed to perform drawing movements from a starting point to a target point which are dis-played on a computer. After completing each movement, the patients will be asked to identify the line they have drawn and to rate how confident they are in identifying the self-drawn line on a scale of 1 - 4 (1 = very unsure, 4 = very sure)
Sensor-based gait and balance analysis | baseline, up to 1 week after intervention, 3, 6, and 12 month follow-up
  movement analysis by wearable movement sensors

CONTACTS AND LOCATIONS:
Overall Officials: Anne Weissbach, MD, Principal Investigator — Institute of Systems Motor Science, University Clinic of Schleswig-Holstein
Locations (2):
- Germany (2):
  - Department of Neurology, University Clinic Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Institute of Systems Motor Science, University Clinic Schleswig-Holstein, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No